CLINICAL TRIAL: NCT04594109
Title: Development of a Tailored Smoking Cessation Program for Individuals With HIV Infection in Washington, D.C.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Jessica Elf, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00022163
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): One-time standard of care in-person behavioral counseling lasting approximately one hour, plus a 30-day supply of nicotine replacement therapy consisting of nicotine patches and nicotine gum (dosage according to current smoking intensity according to manufacturers instructions). The standard of care behavioral counseling was adapted from the current U.S. clinical practice guidelines.
  Interventions: Behavioral: Standard of Care
- Tailored Counseling (Experimental): Participants in the intervention arm were provided a one-time tailored cognitive-behavioral therapy in-person cessation counseling intervention lasting approximately one hour, a 30-day supply of nicotine replacement therapy (consisting of nicotine patches and nicotine gum; dosage according to current smoking intensity according to manufacturers instructions), and a tailored bi-directional text messaging program delivering two messages per day for four weeks. The TI session was adapted from the clinical practice guidelines to include behavioral elements rooted in the minority stress model. The intervention used addressed issues of stress related to HIV stigma, minority status and socioeconomic condition.
  Interventions: Behavioral: Tailored behavioral counseling

INTERVENTIONS:
Behavioral: Tailored behavioral counseling — Participants in the intervention arm were provided a one-time tailored cognitive-behavioral therapy in-person cessation counseling intervention lasting approximately one hour, a 30-day supply of nicotine replacement therapy (consisting of nicotine patches and nicotine gum; dosage according to current smoking intensity according to manufacturers instructions), and a tailored bi-directional text messaging program delivering two messages per day for four weeks. The TI session was adapted from the clinical practice guidelines to include behavioral elements rooted in the minority stress model. The intervention used addressed issues of stress related to HIV stigma, minority status and socioeconomic condition.
  Arms: Tailored Counseling
Behavioral: Standard of Care — One-time standard of care in-person behavioral counseling lasting approximately one hour, plus a 30-day supply of nicotine replacement therapy consisting of nicotine patches and nicotine gum (dosage according to current smoking intensity according to manufacturers instructions). The standard of care behavioral counseling was adapted from the current U.S. clinical practice guidelines.
  Arms: Standard of Care

SUMMARY:
Morbidity and mortality from smoking-related diseases among people living with HIV (PLWH) in the U.S. surpasses that due to HIV itself. Conventional smoking cessation treatments have not demonstrated strong efficacy among PLWH. The investigators conducted a pilot randomized controlled trial (RCT) to evaluate a tailored smoking cessation intervention based on the minority stress model, hypothesizing that behavioral counseling through this lens would enhance cessation. The investigators compared standard of care counseling (SOC) to a tailored intervention (TI) including one face-to-face counseling session incorporating cognitive behavioral therapy to build resilience, and 30 days of 2-way text messaging.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* report being HIV-infected
* be a resident of the Washington, D.C. area
* current, daily smokers of tobacco
* have a confirmed smoking status of 6 parts per million (ppm) or more by using an exhaled carbon monoxide breath monitor
* agree to participate
* be willing to set a quit date within 7 days of baseline assessment.

Exclusion Criteria:

* are currently using smokeless tobacco or electronic cigarettes at least every day
* are currently using nicotine replacement therapy or other smoking cessation treatment
* report being HIV-uninfected
* report having heart disease or high blood pressure not controlled by medication
* are currently in an alcohol treatment program
* are pregnant (exclusion items 4-6 are contraindications of nicotine replacement therapy, which will be provided)
* do not have a primary care provider or HIV care provider to refer to in the event of an adverse reaction to nicotine replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence | 30 day follow-up
  7-day point prevalence plus exhaled breath carbon monoxide < 7 parts per million (ppm)

SECONDARY OUTCOMES:
Cigarettes per day | 30 day follow-up
  Number of cigarettes smoked per day
Exhaled breath carbon monoxide | 30 day follow-up
  Exhaled breath carbon monoxide in parts per million (ppm)
Self-efficacy | 30 day follow-up
  Self-efficacy for smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Elf, PhD MPH, Principal Investigator — Colorado State University
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kierstead EC, Harvey E, Sanchez D, Horn K, Abroms LC, Spielberg F, Stanton CA, Debnam C, Cohn AM, Gray T, Magnus M, Patel M, Niaura R, Elf JL. A pilot randomized controlled trial of a tailored smoking cessation program for people living with HIV in the Washington, D.C. metropolitan area. BMC Res Notes. 2021 Jan 6;14(1):2. doi: 10.1186/s13104-020-05417-3. PMID 33407848